CLINICAL TRIAL: NCT03946397
Title: Impact of Multisensory Hand Massage on the Well-being of Cancer Patients
Acronym: ONCOTACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion issues
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APIRES/2018/IP-01
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory massage (Experimental)
  Interventions: Other: Mulstisensory massage
- Control (No Intervention)

INTERVENTIONS:
Other: Mulstisensory massage — 7 minutes of hand massage followed by multisensory immersion (lights and music) for 23 minutes
  Arms: Multisensory massage

SUMMARY:
The investigators wish to study the impact of a multisensory hand massage on the immediate well-being of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient treated in the oncology department of CHU Nimes for any form of cancer with an EValuation Immédiate du Bien-Etre (EVIBE) score of 3 or lower

Exclusion Criteria:

* The subject is participating in another category I interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient allergic to the massage oil
* Patients with visual or auditory problems
* Patients with an infection resulting in hyperthermia
* Patient with hematoma on the hand
* Patient with dermatological problems or painful areas on the hands
* Patients with an EVIBE score greater than 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Change in well-being following multisensory massage | 30 minutes
  EValuation Immédiate du Bien-Etre (EVIBE) questionnaire: 1-5 pictorial scale with 1 being lowest

SECONDARY OUTCOMES:
Well-being following multisensory massage | 2 hours
  EValuation Immédiate du Bien-Etre (EVIBE) questionnaire: 1-5 pictorial scale with 1 being lowest
Well-being following multisensory massage | 4 hours
  EValuation Immédiate du Bien-Etre (EVIBE) questionnaire: 1-5 pictorial scale with 1 being lowest
Well-being following multisensory massage | 6 hours
  EValuation Immédiate du Bien-Etre (EVIBE) questionnaire: 1-5 pictorial scale with 1 being lowest
Well-being following multisensory massage | 8 hours
  EValuation Immédiate du Bien-Etre (EVIBE) questionnaire: 1-5 pictorial scale with 1 being lowest
Patient anxiety | Immediately prior to treatment
  State Trait Anxiety Inventory (STAI)
Patient anxiety | 30 minutes
  State Trait Anxiety Inventory (STAI)
Patient anxiety | 8 hours
  State Trait Anxiety Inventory (STAI)
Satisfaction of staff performing the multisensory massage | End of inclusions (12 months)
  Custom-built questionnaire; 11 questions on satisfaction at work on a 10-point scale (not at all - enormously)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Houede, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No